CLINICAL TRIAL: NCT01121549
Title: A Non-Interventional Study With Aromasin® As Adjuvant Treatment Of Invasive Early Breast Cancer In Postmenopausal Hormone Receptors Positive Patients Following Of 2-3 Years of Initial Adjuvant Tamoxifen Therapy
Brief Title: A Non-Interventional Study With Aromasin® As Adjuvant Treatment Of Invasive Early Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5991091
Record Dates: First submitted 2010-03-30; First posted 2010-05-12 (Estimated); Results first posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2013-12

CONDITIONS: Invasive Early Breast Cancer
Keywords: Prospective; non-comparative; NIS; 600; postmenopausal; hormone-receptor; positive; EBC; tamoxifen; current medical practice.
MeSH Terms: interventions — exemestane

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aromasin: All patients included in the study
  Interventions: Drug: Aromasin

INTERVENTIONS:
Drug: Aromasin — 25 mg daily continuously
  Other Names: exemestane

SUMMARY:
The IES study (A5991012) investigated 4742 patients treated for 2 to 3 years with tamoxifen, who either continued the same treatment or switched to Aromasin® for a total treatment period of 5 years. Only 65 Romanian patients were enrolled in the IES study. It would therefore appear to be essential to evaluate and confirm the tolerability of Aromasin® and the ways in which it is used on a broader sample of patients and under the standard conditions of use as stipulated in the MA. This Non-Interventional study was designed to address these issues.

DETAILED DESCRIPTION:
This is a prospective, non-comparative, non interventional study (NIS) in four hundred (400) postmenopausal women hormone-receptor positive invasive with early breast cancer, following 2-3 years of initial adjuvant tamoxifen therapy conducted in 60 sites from Romania according to protocol A5991091.The selection of patients based on diagnosis, the attribution of medicinal products and the follow-up of the subjects fall within the current medical practice. A Non-Interventional study is primarily observational in nature. The present Non-interventional Study is performed by medical oncologist and medical oncologist /radiation oncologist who agree to take part in this project. n/a The study was prematurely terminated on August 31th 2012 due to unexpected high rate of patient withdrawal caused by Aromasin reimbursement policy change in Romania; There were no safety issues related to study termination.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal females, defined as one from the next :

  1. Natural menopause >/=1 year,
  2. Surgical ovariectomy,
  3. Chemotherapy-induced amenorrhoea >/=2 years.
* Patients who have had surgical treatment for histological confirmed breast cancer that was non-metastatic at the time of the initial diagnosis.
* Patients who are disease-free after 2 or 3 years of adjuvant tamoxifen treatment.
* Patients whose tumour was estrogen receptor positive (ER+).
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Patients for whom Aromasin® treatment is contraindicated (see SmPC).
* Presence of metastasis or a contra lateral tumour.
* Other adjuvant endocrine therapy.
* Another concomitant antineoplastic treatment
* Participation in a clinical trial with an investigational drug during the 30 days prior to enrolment in the study.
* The patients are not supposed to participate to any other trial during all the study period.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postmenopausal women hormone-receptor positive invasive with early breast cancer, following 2-3 years of initial adjuvant tamoxifen therapy
Sampling Method: Non-Probability Sample
Enrollment: 378 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- Romania (40):
  - Policlinica Judeteana 1 Pitesti - Cabinet oncologie, Piteşti, Argeş
  - Spitalul Judetean de Urgenta Bacau, Bacau, Bacău
  - CMDT MAPN Washington Ambulator oncologie, Bucharest, București
  - Centru D.T. Titan Cabinet oncologie, Bucharest, București
  - Spitalul Judetean de Urgenta Resita Sectia oncologie medicala, Reşiţa, Caraș-Severin County
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta" Cluj Napoca, Cluj-Napoca, Cluj
  - Spitalul Clinic Judetean de Urgenta Cluj, Clinica de Oncologie Medicala si Radioterapie, Cluj-Napoca, Cluj
  - Spitalul Judetean Covasna, Sectia Oncologie medicala, Sfântu Gheorghe, Covasna
  - Spitalul Judetean de Urgenta Targoviste, Târgovişte, Dâmbovița County
  - Spitalulul Judetean de Urgenta Deva, Ambulator oncologie medicala, Hunedoara, Hunedoara County
  - Spitalulul Clinic Judetean de Urgenta Sf. Spiridon, Ambulatoriu de specialitate adulti - Stationar o, Iași, Iaşi
  - Spitalul Clinic Judetean de Urgenta "Sf. Spiridon" Iasi Clinica Oncologie Medicala, Iași, Iaşi
  - Spital Clinic Judetean de Urgenta Oradea, Oradea, Jud. Bihor
  - Spitalul Judeţean Brasov, Brasov, Jud. Brasov
  - Spitalulul Judetean Clinic de Urgenta, Sf. Apostol Andrei, Galati, Jud. Galati
  - Spitalul Judetean Bistrita Nasaud - Sectia Oncologie Medicala, Bistriţa, Jud. Nasaud
  - Spitalul Clinic Judetean de Urgenta Sibiu - Sectia Oncologie Medicala, Sibiu, Jud. Sibiu
  - Spitalul Judetean Drobeta Turnu Severin - Sectie oncologie, Drobeta-Turnu Severin, Mehedinți County
  - Spitalul Judetean Targu Mures, Târgu Mureş, Mureș County
  - Spitalulul Municipal de Urgenta Roman, Roman, Neamț County
  - Spitalul Judetean de Urgenta Slatina, Sectie oncologie, Slatina, Olt
  - Spitalul Municipal Campina Sectia oncologie, Câmpina, Prahova
  - Spitalul Municipal Ploiesti Sectia oncologie, Ploieşti, Prahova
  - Spitalul Municipal Medias Compartimentul Oncologie medicala, Mediaş, Sibiu County
  - Spitalulul Clinic Judetean de Urgenta Sibiu- Sectia Oncologie medicala, Sibiu, Sibiu County
  - Spitalulul Judetean de Urgenta, Sf. Ioan cel Nou, Suceava, Suceava
  - Spitalul Clinic Municipal de Urgenta Timisoara Clinica Oncologie Medicala, Timișoara, Timiș County
  - Spitalul Clinic Municipal Timisoara Sectia oncologie medicala, Timișoara, Timiș County
  - Oncomed Srl, Timișoara, Timiș County
  - Ambulator Spital Colentina, cabinet oncologie, Bucharest
  - Cabinet Oncologie Medicala, Bucharest
  - Ambulator Spital Sf. Pantelimon, cabinet oncolgie, Bucharest
  - Institutul Oncologic "Prof. Dr. Al. Trestioreanu", Bucharest
  - Ambulator Spital Clinic Colţea, cabinet oncologie, Bucharest
  - Policlinica Sf. Ioan Bucuresti, cabinet oncologie, Bucharest
  - Policlinica Theodor Burghele, cabinet oncologie, Bucharest
  - Ambulator Specialitate Cotroceni, cabinet oncolgie, Bucharest
  - Str. Povernei 42, Sector 1, Bucharest
  - Spitalul Clinic de Urgenta, Oradea
  - Spitalul Judetean de Urgenta Targu Jiu, Ambulator Spital - Oncologie medicala, Târgu Jiu

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5991091&StudyName=A%20Non-Interventional%20Study%20With%20Aromasin%AE%20As%20Adjuvant%20Treatment%20Of%20Invasive%20Early%20Breast%20Cancer%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited from Romania.
Groups:
- Exemestane: Participants with 2 to 3 years of initial adjuvant tamoxifen therapy received exemestane (Aromasin) 25 milligram (mg) tablet orally once daily as per local standard of care to complete 5 years of adjuvant hormonal therapy.
Period: Overall Study
Arm/Group | Exemestane
Started | 378
Completed | 31
Not Completed | 347
Not completed — Adverse Event | 10
Not completed — Lack of Efficacy | 11
Not completed — Lost to Follow-up | 12
Not completed — Did not meet entrance criteria | 9
Not completed — Study terminated by sponsor | 197
Not completed — Pregnancy | 1
Not completed — Protocol Violation | 33
Not completed — Withdrawal by Subject | 16
Not completed — Other | 58

BASELINE CHARACTERISTICS:
Arm/Group | Exemestane
Number analyzed (Participants) | 378
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 378
  Male | 0
Number of Participants With Type of Tumor [Number; unit: participants] — Number of participants with different types of tumor such as; ductal carcinoma, lobular carcinoma, invasive ductal carcinoma, invasive lobular carcinoma, papillary carcinoma, medullary carcinoma, mucinous (colloid) carcinoma and others.
  participants
    Ductal Carcinoma | 58
    Lobular Carcinoma | 4
    Invasive Ductal Carcinoma | 246
    Invasive Lobular Carcinoma | 22
    Papillary Carcinoma | 2
    Medullary Carcinoma | 1
    Mucinous (Colloid) Carcinoma | 5
    Other | 24
    Missing/No Response | 16
Number of Participants With Type of Surgery [Number; unit: participants] — Number of participants who had undergone different type of surgeries which included appendicectomy, breast lump removal, cataract operation, cholecystectomy, hysterectomy, intervertebral disc operation, malignant tumor excision, salpingo-oophorectomy bilateral, and splenectomy.
  participants
    Appendicectomy | 6
    Breast lump removal | 1
    Cataract operation | 1
    Cholecystectomy | 17
    Hysterectomy | 3
    Intervertebral disc operation | 1
    Malignant tumor excision | 1
    Salpingo-oophorectomy bilateral | 1
    Splenectomy | 1
Number of Participants With Estrogen Receptor Positive [Number; unit: participants] — Participants whose tumor was estrogen receptor positive are reported.
  participants | 378
Number of Participants With Lymph Node Involvement [Number; unit: participants] | NA — Data for this measure could not be analyzed because case report forms did not provide data for accurate assessment of lymph node involvement.
Number of Participants With Tumor Node Metastasis (TNM) Stage [Number; unit: participants] — TNM was based on size of tumor, if cancer cells had spread to nearby lymph nodes (LN), or distant (to other parts of the body) metastasis had occurred. Stages included: stage 0(no evidence of cancer cells), stage 1(T1N0M0), stage IIA(T0N1M0, T1N1M0, T2N0M0), stage IIB(T2N1M0, T3N0M0), stage IIIA(T0N2M0, T1N2M0, T2N3M0, T3N1orN2M0), stage IIIC(any TN3M0), stage IV(anyT anyNM1), where T0=early form of tumor, T1= <2 centimeter(cm), T2=2-5 cm, T3= >2 cm, T4=large sized tumor, N0=not spread to LN, N1=spread to 1 to 3, N2=spread to 4 to 9, N3=spread >10 axillary LN, M0=no metastasis, M1= Metastasis.
  participants
    Stage I | 64
    Stage IIA | 129
    Stage IIB | 92
    Stage IIIA | 67
    Stage IIIB | 16
    Stage IIIC | 2
    Other | 2
    Missing/No Response | 6
Number of Participants With Histopathological Grade [Number; unit: participants] — The grade of a cancer depends on what the cells look like and the growth-rate. Lower grade indicates a slower-growing cancer and a higher grade indicates a faster-growing one. Grade 1 (resemble normal cells, not growing rapidly), Grade 2 (grow faster than normal cells), Grade 3 and 4 (abnormal cells, grow and spread aggressively).
  participants
    Grade 1 | 62
    Grade 2 | 178
    Grade 3 | 65
    Unknown | 70
    Missing/No Response | 3
Number of Participants With Prior Chemotherapy [Number; unit: participants] | 0
Number of Participants With Prior Radiation Therapy [Number; unit: participants] — A total 271 participants were evaluable for this measure.
  participants | 239

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) by Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs were graded using National Cancer Institute (NCI)/Cancer Therapy Evaluation Program (CTEP) Common Terminology Criteria for Adverse Events version 4.0 (CTCAE,v4.0) as Grade 1 (Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated); Grade 2 (Moderate; minimal, local or noninvasive intervention; limiting age-appropriate instrumental activities of daily living [ADL]); Grade 3 (Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization; disabling; limiting self-care ADL); Grade 4 (Life-threatening; urgent intervention indicated) and Grade 5 (Death related to AE).
Time Frame: Baseline up to 28 days after last dose
Population: Safety analysis set included all participants who had received at least 1 dose of exemestane during the observation period.
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 378
participants
  Grade 1 | 6
  Grade 2 | 8
  Grade 3 | 6
  Grade 4 | 2
  Grade 5 | 0
  Missing or Unknown | 2

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) by Relationship to Study Drug
Description: An AE (all causalities) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to exemestane was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Time Frame: Baseline up to 28 days after last dose
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 378
participants
  AEs (All Causalities) | 24
  SAEs (All Causalities) | 5
  AEs (Treatment Related) | 13
  SAEs (Treatment Related) | 0

3. Secondary Outcome: Number of Missed Exemestane Doses
Time Frame: Week 25, 49, 73, 97, 121, 145
Population: Full analysis set (FAS) included all participants who had received at least 1 dose of exemestane during the observation period. 'N' (number of participants analyzed)=participants evaluable for this measure. n=number of participants evaluable at specified time points. None of the participants were evaluable at Week 145 and hence data not reported.
Measure: Mean (Standard Deviation); unit: missed doses
Arm/Group | Exemestane
Number analyzed (Participants) | 18
missed doses
  Week 25 (n=18) | 4.9 (7.02)
  Week 49 (n=8) | 9.6 (20.40)
  Week 73 (n=5) | 7.6 (12.54)
  Week 97 (n=4) | 12.3 (13.07)
  Week 121 (n=4) | 6.3 (0.50)

4. Secondary Outcome: Number of Participants With Reasons for Discontinuing Exemestane Therapy
Time Frame: Baseline up to Year 3
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 378
participants
  Adverse event | 10
  Insufficient clinical response | 11
  Did not meet entrance criteria | 9
  Lost to follow-up | 12
  No longer willing to participate in study | 16
  Other unspecified | 58
  Protocol violation | 33
  Study terminated by sponsor | 197
  Withdrawn due to pregnancy | 1

5. Secondary Outcome: Number of Participants Who Received Hormonal Therapy or Chemotherapy After Discontinuation of Exemestane Therapy
Time Frame: Baseline up to Year 3
Population: FAS included all participants who had received at least 1 dose of exemestane during the observation period.
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 378
participants
  Received hormonal therapy | 4
  Received chemotherapy | 319
  Received both hormonal and chemotherapy | 1
  No hormonal or chemotherapy received | 34
  Missing or no response | 20

6. Secondary Outcome: Percentage of Participants Who Discontinued the Exemestane Therapy
Time Frame: Baseline up to Year 3
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Exemestane
Number analyzed (Participants) | 378
percentage of participants | 91.8

7. Secondary Outcome: Recurrence-free Survival (RFS)
Description: Recurrence-free survival defined as the time from study inclusion to the first date of documented recurrence, with events defined as: local recurrence, distant recurrence, new primary breast cancer (includes both ipsilateral and contralateral second primaries), or death due to any cause. New primary cancer at sites other than the breast were not considered as recurrence.
Time Frame: Baseline up to Year 3
Population: A subgroup of participants from FAS who had documented recurrence was evaluable for this measure.
Measure: Median (Full Range); unit: weeks
Arm/Group | Exemestane
Number analyzed (Participants) | 14
weeks | 74.357 [27.14 to 133.57]

8. Secondary Outcome: Time to Disease Progression (TTP)
Description: Time to disease progression was defined as the time from inclusion to first local or distant recurrence at any site.
Time Frame: Baseline up to Year 3
Population: Time to disease progression was considered complementary to RFS and hence, was not analyzed.
Arm/Group | Exemestane
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Exemestane
Serious Adverse Events (participants affected / at risk) | 5/378
Other Adverse Events (participants affected / at risk) | 5/378
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=378)
Atrial fibrillation (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Pyelonephritis acute (Infections and infestations) | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=378)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5

LIMITATIONS AND CAVEATS:
The study was prematurely terminated on 31 August 2012 due to unexpected high rate of participant withdrawal caused by Aromasin reimbursement policy change in Romania. There were no safety issues related to study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.